CLINICAL TRIAL: NCT04556318
Title: Study to Identify Differences of Exhaled Breath Components Using Ion Mobility Spectrometry (IMS) in Patients Tested Positive or Negative on SARS-CoV-2
Brief Title: Identification of Differences in Breath Components Detected With IMS in Patients Tested on SARS-CoV-2 (COVID-19)
Status: Completed | Type: Observational
Sponsor: B. Braun Melsungen AG (Industry)
Responsible Party: Sponsor
Other Study IDs: HC-N-H-2004
Record Dates: First submitted 2020-09-18; First posted 2020-09-21 (Actual); Last update posted 2021-07-08 (Actual); Status verified 2021-07

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19 | interventions — Ion Mobility Spectrometry

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Ion Mobility Spectrometry (IMS) — Two breathing gas samples will be taken from each study participant using ion mobility spectrometry with an ultrasound-based spirometer. The total sampling time is 1 minute (at least 5-7 breath takes) following an analysis time of 5-12 minutes.

SUMMARY:
Breath analysis is the evaluation of exhaled air of humans. It aims to get information about the clinical status of a human being by monitoring its volatile organic compounds (VOCs) in exhaled air.

In this feasibility study it is intended to find specific biomarker(s) in exhaled breath indicating an infection with SARS-CoV-2 (severe acute respiratory syndrome coronavirus 2).

ELIGIBILITY:
Inclusion Criteria:

* SARS-CoV-2-Polymerase chain reaction (PCR) test result is available
* Signs or symptoms of any respiratory system infection or Signs or symptoms indicating SARS-CoV-2 infection or Radiological findings suggesting viral lung infection
* Breath test (Study intervention) must be performed within a 2 day time period after latest SARS-CoV-2 PCR

Exclusion Criteria:

* History of SARS-CoV-2 outside the current respiratory episode (known from medical history)
* Participation in another clinical study prior to breath analysis which could influence the result of the breath analysis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with signs or symptoms of any respiratory system infection or signs or symptoms indicating SARS-CoV-2 infection or radiological findings suggesting viral lung infection
Sampling Method: Probability Sample
Enrollment: 396 (Actual)
Dates: Start 2020-09-23 (Actual); Primary Completion 2021-06-11 (Actual); Study Completion 2021-06-11 (Actual)

PRIMARY OUTCOMES:
SARS-CoV-2 related volatile organic compounds (VOC) | 1 hour after breath gas sampling

SECONDARY OUTCOMES:
To compare the SARS-CoV-2 specific VOC with the clinical symptoms of COVID-19 and diagnostic findings | Within 3 days

CONTACTS AND LOCATIONS:
Overall Officials: Christoph Spinner, PD Dr., Principal Investigator — Technical University of Munich, Klinikum rechts der Isar
Locations (2):
- Germany (2):
  - Charité - Universitätsmedizin Berlin, Campus Benjamin Franklin, Berlin
  - Technical University of Munich, Klinikum rechts der Isar, Munich

REFERENCES:
- [Derived] Voit F, Erber J, Feuerherd M, Fries H, Bitterlich N, Diehl-Wiesenecker E, Gladis S, Lieb J, Protzer U, Schneider J, Geisler F, Somasundaram R, Schmid RM, Bauer W, Spinner CD. Rapid point-of-care detection of SARS-CoV-2 infection in exhaled breath using ion mobility spectrometry: a pilot study. Eur J Med Res. 2023 Sep 2;28(1):318. doi: 10.1186/s40001-023-01284-3. PMID 37660038